CLINICAL TRIAL: NCT03861702
Title: A Phase II Study to Evaluate the Efficacy of Liposomal Irinotecan in Combination With Oxaliplatin, Leucovorin, and 5-fluorouracil for Patients With Locally Advanced Pancreatic Carcinoma: Big Ten Cancer Research Consortium BTCRC-GI15-067
Brief Title: Liposomal Irinotecan in Combination With Oxaliplatin, Leucovorin, and 5-fluorouracil for Patients With Locally Advanced Pancreatic Carcinoma:
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nelson Yee (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor-Investigator, Nelson Yee, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GI15-067
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Pancreatic Carcinoma(LAPC)
MeSH Terms: interventions — Folfox protocol; irinotecan sucrosofate

STUDY DESIGN:
Intervention Model Description: This is a phase II, single-arm, open-label, clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFOX + Irinotecan (Experimental): Oxaliplatin 60 mg/m2 Intravenously (IV) over 2 hours
  Liposomal Irinotecan (free base) 50 mg/m2 IV over 90 minutes after completion of oxaliplatin
  Leucovorin 400 mg/m2 IV over 30 minutes after completion of liposomal irinotecan
  5-Fluorouracil 2,400 mg/m2 IV over 46 hours via infusion pump at home
  All drugs administered on day 1 of each 14 day cycle.
  Interventions: Drug: FOLFOX regimen; Drug: Liposomal Irinotecan

INTERVENTIONS:
Drug: FOLFOX regimen — FOLFOX (Oxaliplatin, Leucovorin, 5-Fluorouracil)
Drug: Liposomal Irinotecan — Liposomal Irinotecan
  Other Names: nal-Irinotecan

SUMMARY:
This is a phase II, single-arm, open-label, clinical study to investigate the efficacy and tolerability of a combination of liposomal irinotecan (nal-IRI) with oxaliplatin, leucovorin, and 5-fluorouracil (FOLFOX-nal-IRI) for treatment of patients with locally advanced pancreatic carcinoma (LAPC).

DETAILED DESCRIPTION:
This is a phase II, single-arm, open-label, clinical study to investigate the efficacy and tolerability of a combination of liposomal irinotecan (nal-IRI) with oxaliplatin, leucovorin, and 5-fluorouracil (FOLFOX-nal-IRI) for treatment of patients with locally advanced pancreatic carcinoma (LAPC). Each subject will be screened for eligibility by evaluation including medical history, physical examination, performance status, blood tests, computed tomographic (CT) scans, and electrocardiogram. Within 28 days of screening, the consented subjects will have a central venous access device placed and then start treatment.

For every 2-week cycle of FOLFOX-nal-IRI, each subject will receive nal-IRI (irinotecan free base 50 mg/m2 intravenously over 90 minutes), oxaliplatin (60 mg/m2 intravenously over 2 hours), leucovorin (400 mg/m2 intravenously over 2 hours), and 5-fluorouracil 2,400 mg/m2 intravenously over 46 hours).

Tumor response/surgical assessment will be evaluated after every 4 cycles of treatment with CT scans using RECIST 1.1 criteria. If the tumor becomes surgically resectable and the subject is a surgical candidate as determined by a multidisciplinary team, the subject will undergo surgery (at which point he/she would enter survival follow-up). If the tumor remains unresectable and there is no tumor progression, each subject will be treated up to a total of 12 cycles of FOLFOX-nal-IRI.

Following treatment with 12 cycles of FOLFOX-nal-IRI, if tumor remains unresectable, the subjects may receive further treatment (chemotherapy using the same regimen or of the treating physician's choice, or chemoradiation therapy) or observation as determined by the physician. During the course of treatment, if the subjects develop unacceptable toxicity and/or disease progression, the treatment will be discontinued, and the subjects will be further managed at the discretion of the treating oncologists.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 28 days prior to registration.
* Histological or cytological confirmation of pancreatic carcinoma.
* Measurable disease according to RECIST v1.1 within 28 days prior to registration.
* Previously untreated pancreatic carcinoma considered as locally advanced unresectable according to NCCN guidelines.
* Demonstrate adequate organ function as defined in the table below; All screening labs to be obtained within 14 days prior to initiation of study treatment.

  * Hematological

    * Absolute Neutrophil Count (ANC): >/=1500/uL
    * Hemoglobin (Hgb): >/=8 g/dL with blood transfusion permitted
    * Platelet (Plt): >/=100,000/uL
  * Renal

    * Serum creatinine: </=1.5 x upper limit of normal (ULN) OR
    * Calculated creatinine clearance using the Cockcroft-Gualt formula: >/=50 mL/min for subjects with creatinine levels >1.5 ULN
  * Hepatic

    * Total bilirubin: </=1.5 x ULN (biliary drainage is allowed for biliary obstruction). Patients with Gilbert's syndrome with a total bilirubin </=3.0 x ULN and direct bilirubin within normal limits are permitted
    * Aspartate aminotransferase (AST): </=2.5 x ULN
    * Alanine aminotransferase (ALT): </=2.5 x ULN
    * Albumin: >/=3.0 g/dL
  * Coagulation ---International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT): </=1.5 x ULN unless subject is receiving anticoagulant therapy, as long as PT, INR or PTT is within therapeutic range of intended use of anticoagulants
* Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days of study registration and within 72 hours of Cycle 1 Day 1. NOTE: Female subjects are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Female subjects of childbearing potential and males must be willing to abstain from behaviors that could lead to pregnancy (heterosexual activity, sperm donation, in vitro fertilization, etc.) or to use 2 forms of effective methods of contraception from the time of informed consent until 9 months (females) or 6 months (males) after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study. The subject should be able to understand the purpose and risks of the study and provide a signed and dated informed consent form.

Exclusion Criteria:

* Known hypersensitivity to irinotecan liposome, other liposomal products, oxaliplatin, 5-fluorouracil, leucovorin, or any ingredients in those preparations.
* Pre-existing peripheral neuropathy (Grade 3 or 4) during screening.
* Major surgery within 4 weeks of starting treatment.
* Active uncontrolled cardiac arrhythmia or congestive heart failure (class 3 or 4 as defined by the New York Heart Association Functional Classification); or history of myocardial infarction, unstable angina; or acute coronary syndrome within 6 months prior to enrollment.
* Known history of human immunodeficiency virus (HIV), or hepatic cirrhosis caused by active infection with hepatitis B virus (HBV, as defined by HBsAg positivity or positive DNA). Testing is not required for study entry if there is no clinical suspicion. Note: hepatic cirrhosis caused by other factors (ex. alcoholic cirrhosis) may be considered on a case-by-case basis if, in the opinion of the treating investigator, the disease is unlikely to compromise the subject's safety or put the study outcomes at unnecessary risk.
* Any medical condition, life-threatening illness, or organ dysfunction, which in the investigator's opinion, can compromise the subject's safety or put the study outcomes at unnecessary risk.
* Uncontrolled active systemic infection.
* Concomitant medications that are prohibited in this study and they cannot be switched to alternative medications.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Known additional malignancy that is active and/or progressive requiring treatment within 2 years of screening for this study; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, low-grade prostate cancer, or other cancer for which the subject has been disease-free for at least five years. Additional exceptions could be considered if agreed by sponsor-investigator and site investigator assuming the disease is considered extremely unlikely to confound evaluation of disease status.
* Treatment with any investigational drug within 30 days prior to registration, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Yee, Principal Investigator — Penn State Cancer Institute
Locations (4):
- United States (4):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Rutgers Cancer Institute of new Jersey, New Brunswick, New Jersey
  - Penn State Cancer Institute, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOX + Irinotecan: Oxaliplatin 60 mg/m2 Intravenously (IV) over 2 hours
  Liposomal Irinotecan (free base) 50 mg/m2 IV over 90 minutes after completion of oxaliplatin
  Leucovorin 400 mg/m2 IV over 30 minutes after completion of liposomal irinotecan
  5-Fluorouracil 2,400 mg/m2 IV over 46 hours via infusion pump at home
  All drugs administered on day 1 of each 14 day cycle.
  FOLFOX regimen: FOLFOX (Oxaliplatin, Leucovorin, 5-Fluorouracil)
  Liposomal Irinotecan: Liposomal Irinotecan
Period: Overall Study
Arm/Group | FOLFOX + Irinotecan
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Disease Control Rate (DCR) = CR +PR+SD
Time Frame: Up to 22 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Disease Control Rate was defined as all participants who received at least one dose of trial drug and undergo at least one post-baseline disease assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 26
Percentage of participants | 73

2. Secondary Outcome: Objective Response Rate (ORR) at 8 Weeks
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Overall Response (OR) = CR + PR.
Time Frame: 8 weeks
Population: All participants who have disease assessment at 8 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 25
Percentage of participants | 16

3. Secondary Outcome: Objective Response Rate (ORR) at 16 Weeks
Description: as for outcome 2
Time Frame: 16 weeks
Population: All participants who have disease assessment at 16 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 19
Percentage of participants | 21

4. Secondary Outcome: Objective Response Rate (ORR) at 24 Weeks
Description: as for outcome 2
Time Frame: 24 weeks
Population: All participants who have disease assessment at 24 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 16
Percentage of participants | 25

5. Secondary Outcome: Stable Disease Rate (SDR) at 8 Weeks
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Stable disease rate (SDR) is determined by the proportion of subjects with no progression of disease as defined by RECIST 1.1, at 8 weeks following initiation of FOLFOX-nal-IRI.
Time Frame: 8 Weeks
Population: All participants who have disease assessment at 8 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 25
Percentage of participants | 84

6. Secondary Outcome: Stable Disease Rate (SDR) at 16 Weeks
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Stable disease rate (SDR) as determined by the proportion of subjects with no progression of disease as defined by RECIST 1.1, at 16 weeks following initiation of FOLFOX-nal-IRI.
Time Frame: 16 Weeks
Population: All participants who have disease assessment at 16 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 19
Percentage of participants | 89

7. Secondary Outcome: Stable Disease Rate (SDR) at 24 Weeks
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Stable disease rate (SDR) as determined by the proportion of subjects with no progression of disease as defined by RECIST 1.1, at 24 weeks following initiation of FOLFOX-nal-IRI.
Time Frame: 24 Weeks
Population: All participants who have disease assessment at 24 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 15
Percentage of participants | 80

8. Secondary Outcome: Proportion of Subjects Able to Undergo Surgical Resection
Description: Rate of resectability as determined by the proportion of subjects who undergo surgical resection of tumors.
Time Frame: 12 months
Population: Out of 28 subjects, only 21 subjects had information for surgical resection.
Measure: Number; unit: Proportion of participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 21
Proportion of participants | 0.095

9. Secondary Outcome: Response of Serum CA19-9 Levels
Description: A CA 19-9 test measures the amount of a protein called CA19-9 (cancer antigen 19-9) in a sample of blood. Healthy people can have small amounts of CA 19-9 in their blood. High levels of CA 19-9 are often a sign of pancreatic cancer. Increasing CA 19-9 levels mean the tumor is growing, whether decreasing CA 19-9 levels may mean the tumor is shrinking.
  The Mean of the percentage change from baseline in serum CA19-9 levels associated with best confirmed response (PR, SD, PD) per RECIST 1.1 are reported in the outcome measure data table.
Time Frame: Up to 7 months
Population: All participants who received at least one dose of trial drug, undergo at least one post-baseline disease assessment, and have post-baseline serum CA19-9 information.
Measure: Mean (Standard Deviation); unit: Percentage Change from Baseline
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 25
Percentage Change from Baseline
  Best response: PR: number analyzed (Participants) | 5
  Best response: PR | -69 (37.41)
  Best response: SD: number analyzed (Participants) | 17
  Best response: SD | -41 (40.87)
  Best response: PD: number analyzed (Participants) | 3
  Best response: PD | 31 (8.04)

10. Secondary Outcome: Progression-Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Progression-free survival (PFS) as determined by the time interval from the date of first dose of study drug to first documented disease progression or death from any cause, whichever occurs first.
Time Frame: Up to 22 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Progression-Free Survival was defined as all participants who received at least one dose of trial drug and either undergo at least one post-baseline disease assessment or die before any evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 26
Months | 8.1 [5.19 to 12.1]

11. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as time from the first dose of study drug to date of death from any cause.
Time Frame: Up to 31 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Overall Survival was defined as all participants who received at least one dose of trial drug and either undergo at least one post-baseline disease assessment or die before any evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 26
Months | 18 [11.3 to 22.5]

12. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be assessed to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: Up to 7 months
Population: The analysis population for Adverse Events was defined as all patients who received at least one dose of study treatment regardless of the dosage.
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 28
Participants | 28

13. Secondary Outcome: Quality of Life (QoL) Assessment: Global Health Status (EORTC QLQ-C30)
Description: This secondary outcome measure evaluates overall quality of life using the Global Health Status scale from the EORTC QLQ-C30. Scores range from 0 to 100, with higher scores indicating better global health and quality of life. Mean (SD) scores are reported by assessment period, including only those participants who reached the defined time points (e.g., Cycle 9).
Time Frame: Treatment Cycle 1 (14 days), Treatment Cycle 5 (70 days), Treatment Cycle 9 (126 days), Follow-Up (7 Months)
Population: All participants who reached the specified assessment time points (e.g., Cycle 9) were included in this outcome measure (Total 14 subjects). 13 out of these 14 subjects had information at treatment cycle 1, 12 out of these 14 subjects had information at treatment cycle 5, and 12 out of these 14 subjects had information at Follow-Up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FOLFOX + Irinotecan
Number analyzed (Participants) | 14
score on a scale
  Treatment Cycle 1: number analyzed (Participants) | 13
  Treatment Cycle 1 | 66.7 (26.4)
  Treatment Cycle 5: number analyzed (Participants) | 12
  Treatment Cycle 5 | 69.4 (25.5)
  Treatment Cycle 9 | 68.5 (16.7)
  Follow-Up: number analyzed (Participants) | 12
  Follow-Up | 76.4 (17.0)

ADVERSE EVENTS:
Time Frame: Up to maximum 31 months
Arm/Group | FOLFOX + Irinotecan
All-Cause Mortality (participants affected / at risk) | 13/28
Serious Adverse Events (participants affected / at risk) | 15/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX + Irinotecan (N=28)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
BILIARY TRACT INFECTION (Infections and infestations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 4 (7)
ENTEROCOLITIS (Gastrointestinal disorders) | 2 (3)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
GALLBLADDER INFECTION (Infections and infestations) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 2 (2)
LUNG INFECTION (Infections and infestations) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX + Irinotecan (N=28)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 21 (32)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (3)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 (5)
ANEMIA (Blood and lymphatic system disorders) | 9 (24)
ANOREXIA (Metabolism and nutrition disorders) | 21 (41)
ANOSMIA (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 7 (8)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (7)
BACTEREMIA (Infections and infestations) | 1 (1)
BELCHING (Gastrointestinal disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 1 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2)
BLURRED VISION (Eye disorders) | 2 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 1 (1)
CATARACT (Eye disorders) | 2 (2)
CHILLS (General disorders) | 1 (1)
CHOLESTEROL HIGH (Investigations) | 2 (2)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 3 (3)
CONFUSION (Psychiatric disorders) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 17 (25)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5)
CREATININE INCREASED (Investigations) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4)
DEPRESSION (Psychiatric disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 25 (74)
DIZZINESS (Nervous system disorders) | 9 (10)
DRY EYE (Eye disorders) | 1 (2)
DRY MOUTH (Gastrointestinal disorders) | 4 (5)
DYSESTHESIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 7 (7)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 5 (5)
DYSURIA (Renal and urinary disorders) | 1 (2)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 4 (6)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 3 (3)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 3 (5)
FALL (Injury, poisoning and procedural complications) | 3 (4)
FATIGUE (General disorders) | 22 (55)
FEVER (General disorders) | 3 (9)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 4 (4)
FLOATERS (Eye disorders) | 1 (1)
FLUSHING (Vascular disorders) | 1 (1)
FUNGEMIA (Infections and infestations) | 1 (1)
GALLBLADDER INFECTION (Infections and infestations) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 14 (17)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 10 (11)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 5 (8)
HEART FAILURE (Cardiac disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2)
HERPES SIMPLEX REACTIVATION (Infections and infestations) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 5 (5)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (8)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 6 (6)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 15 (42)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (6)
HYPOKALEMIA (Metabolism and nutrition disorders) | 12 (35)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 4 (6)
HYPONATREMIA (Metabolism and nutrition disorders) | 5 (8)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 4 (6)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2)
ILEUS (Gastrointestinal disorders) | 1 (1)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 1 (3)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 2 (3)
INSOMNIA (Psychiatric disorders) | 10 (11)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 (2)
LOCALIZED EDEMA (General disorders) | 1 (2)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (6)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 5 (8)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 5 (6)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 20 (59)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 3 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 8 (16)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
OBESITY (Metabolism and nutrition disorders) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 1 (3)
PAIN (General disorders) | 3 (6)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PARESTHESIA (Nervous system disorders) | 12 (21)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 13 (29)
PLATELET COUNT DECREASED (Investigations) | 6 (9)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 2 (2)
PSYCHOSIS (Psychiatric disorders) | 1 (1)
RADICULITIS (Nervous system disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
RECTAL FISSURE (Gastrointestinal disorders) | 1 (1)
RECTAL PAIN (Gastrointestinal disorders) | 1 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 3 (3)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SEIZURE (Nervous system disorders) | 1 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (2)
SKIN INFECTION (Infections and infestations) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
SOCIAL CIRCUMSTANCES - OTHER, SPECIFY (Social circumstances) | 1 (1)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (3)
TESTICULAR DISORDER (Reproductive system and breast disorders) | 1 (1)
TESTOSTERONE DEFICIENCY (Endocrine disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 6 (6)
TREMOR (Nervous system disorders) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (2)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 2 (2)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 14 (33)
WEIGHT LOSS (Investigations) | 10 (17)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT03861702/Prot_SAP_000.pdf